CLINICAL TRIAL: NCT01600768
Title: Evaluation of Extended Intravenous of Beta-lactams in the Treatment of Serious Gram-negative Infections in Critically Ill Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200912104M
Record Dates: First submitted 2012-05-16; First posted 2012-05-17 (Estimated); Last update posted 2012-05-17 (Estimated); Status verified 2012-02

CONDITIONS: Gram-Negative Bacterial Infections
Keywords: focus of study
MeSH Terms: conditions — Gram-Negative Bacterial Infections | interventions — beta-Lactams

ARMS (2):
- intermittent infusion (Active Comparator)
  Interventions: Drug: Beta-Lactams
- extended infusion (Experimental)
  Interventions: Drug: Beta-Lactams

INTERVENTIONS:
Drug: Beta-Lactams — infusion time: 30 mins or 1 hr
  Arms: intermittent infusion
Drug: Beta-Lactams — infusion time 4 hrs
  Arms: extended infusion

SUMMARY:
The purpose of this study is to evaluate the PK/PD parameters, safety and efficacy of extended infusion of beta-lactams in intensive care patients who are infected with Gram-negative bacteremia or pneumonia at National Taiwan University Hospital (NTUH).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (> 18 years)
* Admitted on the intensive care unit
* Starting a treatment with beta-lactams antibiotics
* Signed informed consent
* Expected to live > 3 days

Exclusion Criteria:

* renal insufficiency (estimated clearance < 20 ML /MIN)
* renal replacement therapy
* ANC < 1000 103 µl
* pregnancy
* drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-02; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
serum concentrations of beta-lactams | 6 hours
  Determination of serum concentrations of beta-lactams

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Wen Lin, Pharm D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- NTUH, Taipei, Taiwan